CLINICAL TRIAL: NCT04108546
Title: The Effect of Combination of Massage and Electroacupuncture in Patients with Chronic Lumbar Pain. Comparison with the Use of Epidural Analgesia
Brief Title: Massage and Electroacupuncture in Chronic Lumbar Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8/19ης/22-11-2018
Record Dates: First submitted 2019-05-09; First posted 2019-09-30 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Back Pain; Lumbar; Anesthesia, Local; Epidural; Electroacupuncture; Massage
MeSH Terms: conditions — Back Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- massage-electroacupuncture (Experimental): Electroacupuncture will be applied throughout the back of the body, upper limbs and ears.Massage will follow the same paths of acupuncture points respectively
  Interventions: Device: Electroacupuncture device
- Epidural analgesia (Active Comparator): Epidural analgesia will be applied using lidocaine 2%, 1.5 ml, and Dexamethasone 8 mg
  Interventions: Drug: Epidural analgesia

INTERVENTIONS:
Device: Electroacupuncture device — The technical characteristics of the device will be: power supply with alkaline batteries (4 pieces), 6V voltage, 6 independently regulated channels, symmetrical biphasic rectangular pulse, excitation from pen type electrode 0.48mA, with high 0.32mA + / -25% & low 0.16mA +/- 25%. Three preset programs to avoid tolerance effect: program 1) 1-6Hz, program 2) 30-100Hz, program 3) 2-100Hz. Low frequencies (2Hz) cause release of endorphins in the brain and enkephalins in the spinal cord, high frequencies (30-100Hz) cause release of dynorphins in the spinal cord, while medium frequencies (15Hz) cause simultaneous release of endorphin and dynorphin. At low frequencies slow diffuse analgesia is achieved with a long duration of analgesic effect, while at high frequencies rapid local analgesic effect of short duration is achieved.
  Arms: massage-electroacupuncture
Drug: Epidural analgesia — Epidural analgesia with lidocaine 2%, 1.5 ml, and Dexamethasone 8 mg
  Arms: Epidural analgesia

SUMMARY:
The aim of this study is to evaluate and compare in patients with chronic back pain two therapeutic interventions: a) the combination of massage and electroacupuncture; and b) the application of epidural analgesia in pain, functioning-incompetence, quality of life and mood.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from lumbar pain of benign etiology
* Age 20 to 65 years

Exclusion Criteria:

* Ages over 65 or below 20 years
* Neoplasms (benign or malignant etiology)
* Contagious or infectious disease
* Dermopathy
* Pregnancy
* Alcohol or drug use
* Previous use of epidural analgesia
* Systemic opioid use
* Severe heart disease
* Fever for more than one sessions
* Allergy to the oil which will be used and its derivatives
* Thrombi or varicose veins
* Psychiatric disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of pain intensity: NRS | 2 years
  The Numeric Rating Scale will be used to evaluate the pain. The Numeric Pain Rating Scale is a segmented numeric version of the Visual Analog Scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain (0 - no pain, 10 - worst pain).
Assessment of functional status and incompetence in both groups | 2 years
  The Oswestry & Roland-Morris Disability Questionnaire (specific for low-back pain) will be used to assess patient functional status and incompetence
Measurement of health-related quality of life | 2 years
  The SF-36 Health Survey questionnaire will be used. It is a generic measure of health status as opposed to one that targets a specific age, disease, or treatment group. It has three levels: (1) items; (2) eight scales that aggregate 2-10 items each; and (3) two summary measures that aggregate scales. Each item is used in scoring only one scale. Three scales (Physical Functioning, Role-Physical, Bodily Pain) correlate most highly with the physical component and contribute most to the scoring of the Physical Component Summary measure. The mental component correlates most highly with the Mental Health, Role-Emotional, and Social Functioning scales, which also contribute most to the scoring of the Mental Component Summary measure. Three of the scales (Vitality, General Health, and Social Functioning) have noteworthy correlations with both components. The SF-36 has a verbatim content and response choices.
Profile of mood states | 2 years
  The The Profile of Mood States (acronym: POMS) is a standard validated psychological test. This questionnaire will be used to investigate the mood level. It is a questionnaire investigating the mood level and assessing the impact of a program on the patient mood in the short term. The questionnaire consists of 72 adjectives related to mood, which are grouped into 6 factors. The first five factors are negatively rated (high scores correspond to more negative emotions). The sixth factor is scored positively (high scores correspond to higher vitality). Participants are asked to complete these adjectives in a 5-point Likert-type scale ranging from "not at all" (0) to "extremely" (4).

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - University Hospital of Larisa, Department of Anesthesiology, Larissa, Thessaly
  - University Hospital of Larissa, Larissa, Thessaly

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andrianakos A, Trontzas P, Christoyannis F, Dantis P, Voudouris C, Georgountzos A, Kaziolas G, Vafiadou E, Pantelidou K, Karamitsos D, Kontelis L, Krachtis P, Nikolia Z, Kaskani E, Tavaniotou E, Antoniades C, Karanikolas G, Kontoyanni A; ESORDIG Study. Prevalence of rheumatic diseases in Greece: a cross-sectional population based epidemiological study. The ESORDIG Study. J Rheumatol. 2003 Jul;30(7):1589-601. PMID 12858464
- [Background] Diatchenko L, Anderson AD, Slade GD, Fillingim RB, Shabalina SA, Higgins TJ, Sama S, Belfer I, Goldman D, Max MB, Weir BS, Maixner W. Three major haplotypes of the beta2 adrenergic receptor define psychological profile, blood pressure, and the risk for development of a common musculoskeletal pain disorder. Am J Med Genet B Neuropsychiatr Genet. 2006 Jul 5;141B(5):449-62. doi: 10.1002/ajmg.b.30324. PMID 16741943
- [Background] Diego MA, Field T, Sanders C, Hernandez-Reif M. Massage therapy of moderate and light pressure and vibrator effects on EEG and heart rate. Int J Neurosci. 2004 Jan;114(1):31-44. doi: 10.1080/00207450490249446. PMID 14660065
- [Background] Fang JQ, Du JY, Fang JF, Xiao T, Le XQ, Pan NF, Yu J, Liu BY. Parameter-specific analgesic effects of electroacupuncture mediated by degree of regulation TRPV1 and P2X3 in inflammatory pain in rats. Life Sci. 2018 May 1;200:69-80. doi: 10.1016/j.lfs.2018.03.028. Epub 2018 Mar 14. PMID 29550358
- [Background] Richardson JC, Ong BN, Sim J. Experiencing and controlling time in everyday life with chronic widespread pain: a qualitative study. BMC Musculoskelet Disord. 2008 Jan 11;9:3. doi: 10.1186/1471-2474-9-3. PMID 18190693
- [Background] Yamashita H, Tsukayama H, Tanno Y, Nishijo K. Adverse events in acupuncture and moxibustion treatment: a six-year survey at a national clinic in Japan. J Altern Complement Med. 1999 Jun;5(3):229-36. doi: 10.1089/acm.1999.5.229. PMID 10381246